CLINICAL TRIAL: NCT03171922
Title: Effects of Internet-based Diet Plus Online Dietary Coach Compared With in Person Clinic Visit Approach on Weight Loss in Healthy Obese Women in a Weight-loss Program: a Randomized Clinical Trial
Brief Title: Effects of Internet-based Diet Plus Online Dietary Coach Compared With in Person Clinic Visit Approach on Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novindiet Clinic (Other)
Collaborators: University of Nottingham (Other); Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-206
Record Dates: First submitted 2017-05-27; First posted 2017-05-31 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-01

CONDITIONS: Obesity; Overweight
Keywords: weight loss; internet-based diet; online dietary coach; clinic visit approach; Diet
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet Diet (Experimental): Internet Diet group have online dietary coach every 2 weeks
  Interventions: Behavioral: Internet Diet
- Clinic Diet (Experimental): clinic visit based weight loss diet program group who have every 2 weeks visit at clinic.
  Interventions: Behavioral: Clinic Diet

INTERVENTIONS:
Behavioral: Internet Diet — ID group have online dietary coach every 2 weeks
  Other Names: ID
  Arms: Internet Diet
Behavioral: Clinic Diet — CD group have every 2 weeks visit at clinic
  Other Names: CD
  Arms: Clinic Diet

SUMMARY:
The purpose of this study is to examine the efficacy of an internet based diet plus a regular dedicated dietary coach (ID group) versus clinic visit based weight loss program (CD group) on weight loss in obese and overweight female adults.

ELIGIBILITY:
Inclusion Criteria:

* Must be female
* Must be 18-45 years of age.
* Must have Body mass index (BMI) between 27-35 kg/ m².
* Must be able to have moderate exercise.
* Must be interested to have weight loss.
* Have access to a personal computer and the Internet

Exclusion Criteria:

* Pregnancy or lactation during the previous 6 months, or planned pregnancy in the next six months.
* Taking medications that could affect metabolism or change body weight.
* Report heart problems, chest pain, and cancer within the last five years.
* Smoking
* Menopause
* Diagnosis of any chronic disease such as fatty liver, cancer, chemo/radio therapy, heart disease, immune compromised conditions, abnormal thyroid hormone level.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2018-09-29 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Weight | 1year
  kg

SECONDARY OUTCOMES:
Waist circumference | 1year
  cm
fasting blood glucoses | 1year
  mmol/l
fasting insulin level | 1year
  mU/l
HbA1c | 1year
  Score
HOMA-IR | 1year
  percentage (%)
lipid profiles | 1year
  mmol/l
liver function tests | 1year
  U/l

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - NovinDiet Clinic, Tehran
  - NovinDiet Clinic, Tehrān

IPD SHARING:
Plan to Share IPD: Undecided